CLINICAL TRIAL: NCT02622035
Title: New Technology and Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 160026; 16-HG-0026
Record Dates: First submitted 2015-12-03; First posted 2015-12-04 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Child Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1 (Experimental): Gain frame; Anger
  Interventions: Behavioral: Provision of information; Behavioral: Emotion induction
- 1b (Experimental): high visual perceptual load high interactive
  Interventions: Behavioral: visual perceptual load
- 2 (Experimental): Gain frame; Fear
  Interventions: Behavioral: Provision of information; Behavioral: Emotion induction
- 2b (Experimental): high visual perceptual load
  Interventions: Behavioral: visual perceptual load
- 3 (Experimental): Loss frame; Anger
  Interventions: Behavioral: Provision of information; Behavioral: Emotion induction
- 3b (Experimental): low visual perceptual load
  Interventions: Behavioral: visual perceptual load
- 4 (Experimental): Loss frame; Fear
  Interventions: Behavioral: Provision of information; Behavioral: Emotion induction

INTERVENTIONS:
Behavioral: Provision of information — Information about fruit and vegetable feeding for children framed in gain vs. loss manner
  Arms: 1; 2; 3; 4
Behavioral: Emotion induction — Film clip designed to induce anger or fear
  Arms: 1; 2; 3; 4
Behavioral: visual perceptual load — visual and interactivity-based load of virtual reality buffet environment
  Arms: 1b; 2b; 3b

SUMMARY:
Background:

We are involved in testing new behavioral science methods and measures for future research projects. In the course of these evaluations, we will also test research questions related to parents psychological experiences and how these relate to the responses they have when they encounter different types of communication about child health. We are testing multiple research questions in the course of this research.

Objective:

- To learn about technologies and approaches to use in future research studies.

Eligibility:

- Parents (fathers and mothers) of children between the ages of 3-7.

Design:

As part of the main study, participants will do four tasks:

Task 1: Before participants arrive for an in-person visit, they will answer questions online about themselves, their child, and their thoughts and opinions related to health.

Task 2: At the in-person visit, participants will watch a short scene from a movie and answer some questions

Task 3: At the in-person visit, participants will read information about a child health topic and answer questions

Task 4: At the in-person visit, participants will use a virtual reality-based buffet restaurant simulation to make hypothetical food choices for their child...

DETAILED DESCRIPTION:
Background:

We are involved in testing new behavioral science methods and measures for future research projects. In the course of these evaluations, we will also test research questions related to parents psychological experiences and how these relate to the responses they have when they encounter different types of communication about child health. We are testing multiple research questions in the course of this research.

Objective:

- To learn about technologies and approaches to use in future research studies.

Eligibility:

- Parents (fathers and mothers) of children between the ages of 3-7.

Design:

As part of the main study, participants will do four tasks:

Task 1: Before participants arrive for an in-person visit, they will answer questions online about themselves, their child, and their thoughts and opinions related to health.

Task 2: At the in-person visit, participants will watch a short scene from a movie and answer some questions

Task 3: At the in-person visit, participants will read information about a child health topic and answer questions

Task 4: At the in-person visit, participants will use a virtual reality-based buffet restaurant simulation to make hypothetical food choices for their child

ELIGIBILITY:
* INCLUSION CRITERIA - MAIN TRIAL
* All participants in the main trial will be healthy adult parents 18 years and older
* Inclusion criteria include:

  1. being the parent of a biological child who is between 4 and 7 years old with no major allergies or dietary-related health conditions;
  2. having some responsibility for child s dietary intake ;
  3. having the ability to read, write, and converse in English;
  4. being able to come to the NIH Clinical Center for one visit.

EXCLUSION CRITERIA - MAIN TRIAL

* Exclusion criteria include:

  1. having received information about the study purpose;
  2. being an NHGRI employee;
  3. being from a family wherein another household member or co-parent of a biological child has already participated or is scheduled to participate.

     EXCLUSION CRITERIA - VIRTUAL REALITY
* Exclusion criteria related to use of the virtual reality environment include:

  1. having a medical susceptibility to dizziness, disorientation or nausea;
  2. having a seizure disorder or epilepsy;
  3. having a high propensity for motion sickness;
  4. lacking freedom of movement;
  5. known pregnancy;
  6. low, uncorrected vision and hearing.

INCLUSION CRITERIA - PILOT

* Participants in the Pilot test will be healthy adult parents 18 years and older.
* Inclusion criteria include:

  1. being the parent of a biological child who is between 3 and 7 years old with no major allergies or dietary-related health conditions, but only for the first 10 participants;
  2. having the ability to read, write, and converse in English;
  3. being able to come to the NIH Clinical Center for one visit.

EXCLUSION CRITERIA - PILOT

1. having received information about the study purpose;
2. being an NHGRI employee;
3. low, uncorrected vision and hearing.

INCLUSION CRITERIA - BUFFET SERVING EVALUATION

* Participants in the secondary Buffet Serving Evaluation will be healthy adult parents 18 years and older
* Inclusion criteria include:

  1. being the parent of a biological child who is between 3 and 7 years old with no major allergies or dietary-related health conditions;
  2. having some responsibility for child s dietary intake ;
  3. having the ability to read, write, and converse in English;
  4. being able to come to the NIH Clinical Center for one visit.

EXCLUSION CRITERIA - BUFFET SERVING EVALUATION (MAIN)

1. being an NHGRI employee;
2. being from a family wherein another household member or co-parent of a biological child has already participated or is scheduled to participate.

EXCLUSION CRITERIA - BUFFET SERVING EVALUATION (VIRTUAL REALITY)

* Exclusion criteria related to use of the virtual reality environment include:

  1. having a medical susceptibility to dizziness, disorientation or nausea;
  2. having a seizure disorder or epilepsy;
  3. having a high propensity for motion sickness;
  4. lacking freedom of movement;
  5. known pregnancy;
  6. low, uncorrected vision and hearing.

     INCLUSION CRITERIA- OLFACTORY AWARENESS TEST:
* Participants in the Olfactory Awareness Test will be healthy adults between the ages of 18 and 59

Inclusion criteria include:

1. Having the ability to read, write and converse in English
2. Able to come to the clinical center for on visit.

We may also include the following inclusion criteria:

1. Being the parent of a biological child who is between 3 and 7 years old with no major allergies or dietary-related health conditions
2. Having some responsibility for child s dietary intake; however, if we encounter recruitment difficulties, we may instead sample nonparent participants who are of the same general age range as parents who participated in our past studies using the virtual buffet. For the pilot test, we will sample non-parents in the age range of past parent participants

EXCLUSION CRITERIA-OLFACTORY AWRAENESS TEST:

1. Being an NHGRI employee;
2. Having participated in the Parents TAKE study conducted previously in this lab.

Exclusion criteria related to use of the virtual reality environment include:

1. Having a medical susceptibility to dizziness, disorientation or nausea;
2. Having a seizure disorder or epilepsy;
3. Having a high propensity for motion sickness;
4. Lacking freedom of movement;
5. Known pregnancy;
6. Weak, uncorrected vision, hearing, and/or smell. No adults older than age 59 will be able to participate in this study because older adults tend to experience a decline in olfactory function

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Exhibited emotion, Feeding decisions, self-reported attitudes, beliefs and intentions; perceptual responses | At lab visit
  feeding behavior and self-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Susan Persky, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data set is not currently deidentified and participants were not consented for data sharing.

REFERENCES:
- [Derived] Persky S, Ferrer RA, Klein WMP, Goldring MR, Cohen RW, Kistler WD, Yaremych HE, Bouhlal S. Effects of Fruit and Vegetable Feeding Messages on Mothers and Fathers: Interactions Between Emotional State and Health Message Framing. Ann Behav Med. 2019 Aug 16;53(9):789-800. doi: 10.1093/abm/kay088. PMID 30395145
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-HG-0026.html